CLINICAL TRIAL: NCT04006288
Title: Switching From Standard of Care Dual Antiplatelet Treatment (DAPT) Regimens With Aspirin Plus a P2Y12 Inhibitor to Dual Pathway Inhibition (DPI) With Low-dose Rivaroxaban in Adjunct to Aspirin in Patients With Coronary Artery Disease: The Switching Anti-Platelet and Anti-Coagulant Therapy (SWAP-AC) Study
Brief Title: Switching From DAPT to Dual Pathway Inhibition With Low-dose Rivaroxaban in Adjunct to Aspirin in Patients With Coronary Artery Disease
Acronym: SWAP-AC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS-RIVA02
Record Dates: First submitted 2019-06-25; First posted 2019-07-05 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease
Keywords: dual antiplatelet therapy; rivaroxaban; pharmacodynamic
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Prasugrel Hydrochloride; Ticagrelor; Aspirin; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Patients treated with either aspirin (81mg/qd) plus clopidogrel, aspirin (81mg/qd) plus ticagrelor (90mg/bid), or aspirin (81mg/qd) plus prasugrel (10mg/bid) will be identified. Each cohort will be randomized 1:1 to either maintain DAPT or to DPI. DPI consists in treatment with aspirin (81mg/qd) plus rivaroxaban (2.5mg/bid). Patients randomized to DAPT will continue their guideline recommended DAPT regimens.
Masking Description: laboratory personnel running pharmacodynamic testing will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Aspirin and clopidogrel (Active Comparator): aspirin 81 mg/qd plus clopidogrel 75mg/qd for 30 days
  Interventions: Drug: Clopidogrel; Drug: aspirin
- Aspirin and rivaroxaban from aspirin and clopidogrel (Experimental): aspirin 81mg/qd plus rivaroxaban 2.5mg/bid for 30 days
  Interventions: Drug: aspirin; Drug: rivaroxaban
- Aspirin and prasugrel (Active Comparator): aspirin 81 mg/qd plus prasugrel 10mg/qd for 30 days
  Interventions: Drug: Prasugrel; Drug: aspirin
- Aspirin and rivaroxaban from aspirin and prasugrel (Experimental): aspirin 81mg/qd plus rivaroxaban 2.5mg/bid for 30 days
  Interventions: Drug: aspirin; Drug: rivaroxaban
- Aspirin and ticagrelor (Active Comparator): aspirin 81 mg/qd plus ticagrelor 60mg/bid for 30 days
  Interventions: Drug: ticagrelor; Drug: aspirin
- Aspirin and rivaroxaban from aspirin and ticagrelor (Experimental): aspirin 81mg/qd plus rivaroxaban 2.5mg/bid for 30 days
  Interventions: Drug: aspirin; Drug: rivaroxaban

INTERVENTIONS:
Drug: Clopidogrel — Patients on aspirin and plavix will be randomized to either continue with aspirin and plavix or to switch to aspirin and rivaroxaban
  Other Names: Plavix
  Arms: Aspirin and clopidogrel
Drug: Prasugrel — Patients on aspirin and prasugrel will be randomized to either continue with aspirin and prasugrel or to switch to aspirin and rivaroxaban
  Other Names: Effient
  Arms: Aspirin and prasugrel
Drug: ticagrelor — Patients on aspirin and ticagrelor will be randomized to either continue with aspirin and ticagrelor or to switch to aspirin and rivaroxaban
  Other Names: brilinta
  Arms: Aspirin and ticagrelor
Drug: aspirin — all patients will remain on aspirin
Drug: rivaroxaban — Patients on DAPT will be randomized to either continue with DAPT or to switch to aspirin and rivaroxaban
  Other Names: xarelto
  Arms: Aspirin and rivaroxaban from aspirin and clopidogrel; Aspirin and rivaroxaban from aspirin and prasugrel; Aspirin and rivaroxaban from aspirin and ticagrelor

SUMMARY:
Recent studies indicate that anti-factor-Xa inhibition with low-dose rivaroxaban may have a role in the reduction of ischemic recurrences in patients with atherosclerotic disease manifestations. The objectives of this investigation are to assess the feasibility of switching from a DAPT to DPI regimen and to compare the pharmacodynamic profiles of these treatment regimens. This will be a prospective study conducted in cohorts of patients with CAD on treatment per standard of care with DAPT. Patients will be randomized to either maintain DAPT or to DPI. DPI consists in treatment with aspirin (81mg/qd) plus rivaroxaban (2.5mg/bid).

DETAILED DESCRIPTION:
Recent studies indicate that anti-factor-Xa inhibition with low-dose rivaroxaban may have a role in the reduction of ischemic recurrences in patients with atherosclerotic disease manifestations. In the COMPASS trial, patients with stable coronary or peripheral artery disease and no indication for oral anticoagulation or dual antiplatelet therapy (DAPT) were randomized to rivaroxaban 2.5 mg bid in combination with aspirin, rivaroxaban 5 mg bid monotherapy or aspirin monotherapy. The study showed a significant 24% relative reduction in ischemic outcomes with rivaroxaban 2.5 mg bid plus aspirin combination strategy compared with aspirin alone. These observations have raised practical considerations on how to implement the results of the COMPASS trial in clinical practice particularly for patients who are completing a minimum duration of DAPT and contemplating between continuing with a DAPT regimen versus switching to a dual pathway inhibition (DPI) regimen with aspirin plus rivaroxaban. Therefore, the objectives of this investigation are to assess the feasibility of switching from a DAPT to DPI regimen and to compare the pharmacodynamic profiles of these treatment regimens. This will be a prospective study conducted in cohorts of patients with CAD on treatment per standard of care with DAPT. Patients will be randomized to either maintain DAPT or to DPI. DPI consists in treatment with aspirin (81mg/qd) plus rivaroxaban (2.5mg/bid).

ELIGIBILITY:
Inclusion criteria:

* Willing and able to provide written informed consent
* Above 18 years of age
* Have known CAD and have completed their required duration of standard of care DAPT (aspirin in combination with either clopidogrel, prasugrel, or ticagrelor) and still be on treatment:

  * ≥ 6 months after an elective PCI
  * ≥ 12 months after experiencing an ACS (irrespective of revascularization at the time of ACS; thus patients treated by PCI, CABG, or medically managed can be considered)

Exclusion criteria:

* Deemed to be at high risk of bleeding, active bleeding or history of major bleeding Stroke within 1 month or any history of hemorrhagic or lacunar stroke
* Estimated glomerular filtration rate <15 mL/min by MDRD equation
* Need for dual antiplatelet therapy, other non-aspirin antiplatelet therapy, or oral anticoagulant therapy
* Known non-cardiovascular disease that is associated with poor prognosis (e.g., metastatic cancer) or that increases the risk of an adverse reaction to study interventions.
* History of hypersensitivity or known contraindication for rivaroxaban.
* Systemic treatment with strong inhibitors of both CYP 3A4 and p-glycoprotein (e.g., systemic azole antimycotics, such as ketoconazole, and human immunodeficiency virus [HIV]-protease inhibitors, such as ritonavir), or strong inducers of CYP 3A4, i.e.

rifampicin, rifabutin, phenobarbital, phenytoin, and carbamazepine

* Any known hepatic disease associated with coagulopathy
* Subjects who are pregnant, breastfeeding, or are of childbearing potential, and sexually active and not practicing an effective method of birth control (e.g. surgically sterile, prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, contraceptive patch, male partner sterilization)
* Concomitant participation in another study with investigational drug
* Known contraindication to any study related procedures
* Hemoglobin ≤9 mg/dL
* Platelet count <80x106/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ortega-Paz L, Franchi F, Rollini F, Galli M, Been L, Ghanem G, Shalhoub A, Ossi T, Rivas A, Zhou X, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Jennings LK, Angiolillo DJ. Switching from Dual Antiplatelet Therapy with Aspirin Plus a P2Y12 Inhibitor to Dual Pathway Inhibition with Aspirin Plus Vascular-Dose Rivaroxaban: The Switching Anti-Platelet and Anti-Coagulant Therapy (SWAP-AC) Study. Thromb Haemost. 2024 Mar;124(3):263-273. doi: 10.1055/a-2098-6639. Epub 2023 May 24. PMID 37224883

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients treated with either aspirin (81mg/qd) plus clopidogrel, aspirin (81mg/qd) plus ticagrelor (90mg/bid), or aspirin (81mg/qd) plus prasugrel (10mg/bid) were identified. Each cohort was randomized 1:1 to either maintain DAPT or to DPI. DPI consists in treatment with aspirin (81mg/qd) plus rivaroxaban (2.5mg/bid). Patients randomized to DAPT will continue their guideline recommended DAPT regimens.
Period: Overall Study
Arm/Group | Aspirin and Clopidogrel | Aspirin and Rivaroxaban From Aspirin and Clopidogrel | Aspirin and Prasugrel | Aspirin and Rivaroxaban From Aspirin and Prasugrel | Aspirin and Ticagrelor | Aspirin and Rivaroxaban From Aspirin and Ticagrelor
Started | 15 | 15 | 15 | 15 | 15 | 15
Completed | 14 | 14 | 15 | 15 | 15 | 15
Not Completed | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin and Clopidogrel | Aspirin and Rivaroxaban From Aspirin and Clopidogrel | Aspirin and Prasugrel | Aspirin and Rivaroxaban From Aspirin and Prasugrel | Aspirin and Ticagrelor | Aspirin and Rivaroxaban From Aspirin and Ticagrelor | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.9) | 64.1 (7.2) | 61.1 (6.6) | 61.1 (9.0) | 56.5 (8.8) | 60.9 (9.4) | 61.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 12 | 12 | 8 | 11 | 60
  Male | 8 | 5 | 3 | 3 | 7 | 4 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 4 | 3 | 5 | 4 | 28
  White | 9 | 9 | 10 | 12 | 10 | 11 | 61
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 15 | 15 | 15 | 15 | 90
Diabetes mellitus [Count of Participants; unit: Participants] | 11 | 9 | 10 | 5 | 12 | 7 | 54
Previous percutaneous coronary intervention [Count of Participants; unit: Participants] | 13 | 12 | 15 | 15 | 15 | 15 | 85

OUTCOME MEASURES:

1. Primary Outcome: Maximal Platelet Aggregation (MPA%) by Light Transmittance Aggregometry (LTA)
Description: The primary end point of this study will be the comparison of MPA% measured by LTA using the CATF cocktail as agonist between DAPT and low-dose rivaroxaban plus aspirin for each DAPT regimen
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: percentage of MPA
Arm/Group | Aspirin and Clopidogrel | Aspirin and Rivaroxaban From Aspirin and Clopidogrel | Aspirin and Prasugrel | Aspirin and Rivaroxaban From Aspirin and Prasugrel | Aspirin and Ticagrelor | Aspirin and Rivaroxaban From Aspirin and Ticagrelor
Number analyzed (Participants) | 14 | 14 | 15 | 15 | 15 | 15
percentage of MPA | 27 [17 to 50] | 53 [43 to 66] | 20 [4 to 37] | 4 [0 to 17] | 15 [1 to 33] | 20 [6 to 50]

ADVERSE EVENTS:
Time Frame: At 30 days.
Description: Ischemic and bleeding according to the Bleeding Academic Research Consortium (BARC) definition.
Arm/Group | Aspirin and Clopidogrel | Aspirin and Rivaroxaban From Aspirin and Clopidogrel | Aspirin and Prasugrel | Aspirin and Rivaroxaban From Aspirin and Prasugrel | Aspirin and Ticagrelor | Aspirin and Rivaroxaban From Aspirin and Ticagrelor
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15 | 0/15 | 0/15 | 0/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin and Clopidogrel (N=15) | Aspirin and Rivaroxaban From Aspirin and Clopidogrel (N=15) | Aspirin and Prasugrel (N=15) | Aspirin and Rivaroxaban From Aspirin and Prasugrel (N=15) | Aspirin and Ticagrelor (N=15) | Aspirin and Rivaroxaban From Aspirin and Ticagrelor (N=15)
Bleeding (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT04006288/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT04006288/ICF_001.pdf